CLINICAL TRIAL: NCT02040311
Title: A Multicenter Randomized, Double-blind, Placebo-controlled, Parallel Group Study of the Efficacy and Safety of Topiramate in Weight Loss Maintenance in Obese Subjects Following Participation in an Intensive, Non-pharmacologic Weight Loss Program
Brief Title: Topiramate: Long-Term Maintenance of Weight Loss Induced by Low-Calorie Diet in Obese Subjects
Acronym: TOBES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated early as sponsor wanted to develop an improved formulation.
Sponsor: University of Copenhagen (Other)
Collaborators: R W Johnson Pharmaceutical Research Institute (Industry)
Responsible Party: Principal Investigator, Arne Astrup, ph.D, M.D., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRI/TOP-INT-35
Record Dates: First submitted 2014-01-07; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topiramate 96 mg daily (Experimental)
  Interventions: Drug: Topiramate 96 mg daily
- Topiramate 192 mg daily (Experimental)
  Interventions: Drug: Topiramate 192 mg daily
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate 96 mg daily
  Arms: Topiramate 96 mg daily
Drug: Topiramate 192 mg daily
  Arms: Topiramate 192 mg daily
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of topiramate (96 mg or 192 mg daily) as compared to placebo in maintaining weight loss in obese subjects who participated in an eight week intensive non-pharmacologic weight loss program.

The primary efficacy endpoint will be the percent change in body weight from enrollment visit to week 60.

DETAILED DESCRIPTION:
The study was a randomized, double-blind, placebo-controlled, parallel-group, multicenter trial. It was originally designed to last a total of 74 weeks: an 8 week non.pharmacologic low-calorie (800 to 1000 kcl/d) weight loss run-in phase, an 8 week titration phase, 52 week maintenance phase, and 6 week drug taper and follow up phase.

ELIGIBILITY:
Inclusion Criteria:

* Read and signed the informed consent form after the nature of the study has been fully explained
* 18 to 75 years og age at enrollment
* subjects must have either:

  1. A body mass index BMI ≥ 33 kg/m*m and < 50 kg/m*m, or
  2. A BMI ≥ 30 kg/m*m < 50 kg/m*m if any of the following established co-morbidities are present:

Controlled hypertension or dyslipidemia. Anti-hypertensive and hypo-lipidemic medication should have been at a stable dose for at least two months prior to enrollment. If subjects are clinically diagnosed with any of these conditions as a result of enrollment assessments, they can only continue in the enrollment phase if in the clinical judgment of the investigator initiation of anti-hypertensive or hypo-lipidemic therapy is not required.

* Subjects diagnosed with type 2 diabetes by means of OGTT at enrollment visit and not requiring anti diabetic therapy according to the clinical judgement of the investigator.
* Stable weight (varying to more than 3 kg) for at least 3 months prior to enrollment.
* Female subjects must be post menopausal for at least a year or surgically incapable of childbearing, practicing abstinence an acceptable method of birth control. If a female subject of child bearing potential is practicing an acceptable method of birth control, she must have had a negative urine pregnancy test at enrollment, as well as at baseline, prior to receiving study drug.

Randomization criteria

1. Weight reduction of≥ 8% of enrollment body weight at the randomization visit;
2. Subjects must have either:

2a) A BMI ≥ 30 kg/m*m and < 50 kg/m*m, or 2b) A BMI ≥ 27 kg/m*m and < 50 kg/m*m if any of the following established co-morbidities are present: controlled hypertension or dyslipidemia.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in the study.

* Prior exposure or known contraindication or hypersensitivity to topiramate;
* Exposure to any other experimental drug or device within 30 days prior to enrollment;
* Pregnancy or nursing or subjects who plan to become pregnant during the study;
* An established diagnosis of diabetes prior to study enrollment;
* History or evidence of clinically significant hepatic disease;
* Evidence of renal impairment;
* Significant cardiovascular disease;
* Uncontrolled hypertension 180 / 100 mmHg
* Hypertensive subjects on medications must have been on the same dose of the same hypertensive medication for at least 2 months;
* Uncontrolled thyroid disease including hyper- or hypothyroidism or an abnormal TSH-level;
* A history of obesity with a known cause e.g. Cushings disease;
* A history or family history (first degree relatives) of kidney stones;
* Previous gastric restrictive surgery or other surgical procedures to cause weight loss, including liposuction;
* History of gluten or non-gluten induced enteropathy;
* Clinically significant lactose intolerance, in the opinion of the investigator;
* Malignancy or with a history of malignancy within 5 years prior to enrollment, other than basal cell carcinomas of the skin;
* History og seizures or significant CNS disorders;
* History of significant psychiatric disorders including schizophrenia, psychosis and major affective disorders;
* History of anorexia nervosa, bulimia og binge eating disorder;
* A significant change in smoking habit within 2 months of the enrollment visit, in the opinion of the investigator;
* History of drug or alcohol abuse within the previous 2 years;
* Positive results on any urine drug screen at enrollment;
* Use of any weight loss preparations within 30 days prior to enrollment;
* Use of any systemic corticosteroids within 30 days prior to enrollment;
* Clinically significant hematological or immunological disorder;
* Currently receiving psychotropic medications, except episodic use of certain medications;
* Receiving any excluded medication, depending on episodic or chronic use;
* Any significant condition that, in the opinion of the investigator, could interfere with the subjects participation or compliance in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2000-08; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
weight loss | 60 weeks

SECONDARY OUTCOMES:
blood lipids | 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arne V Astrup, phD.MD, Principal Investigator — Department of Human Nutrition
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark